CLINICAL TRIAL: NCT04720313
Title: A Phase 1 Dose Escalation and Safety Study of NXC-201 (formerly HBI0101) CART in BCMA-Expressing Multiple Myeloma Patients
Brief Title: NXC-201 (formerly HBI0101) Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Nexcella Inc. (Industry)
Responsible Party: Principal Investigator, Polina Stepensky, Professor, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOH_2020-12-22_009584
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Dose Escalation and Safety

STUDY DESIGN:
Intervention Model Description: Multiple Myeloma and AL amyloidosis Patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CART BCMA (Experimental): The dose escalation phase (Part A) will include the following doses of CAR-positive (CAR+) T cells: 150×10^6, 450×10^6, 800×10^6 or 1200 ×10^6 The expansion phase (Part B) will include a dose between 450×10^6 to 800×10^6 CAR-positive (CAR+) T cells
  Interventions: Drug: NXC-201 (formerly HBI0101)

INTERVENTIONS:
Drug: NXC-201 (formerly HBI0101) — NXC-201 (formerly HBI0101) CART is defined as autologous T cells transduced ex-vivo with anti-BCMA CAR retroviral vector encoding the chimeric antigen receptor (CAR) targeted to human BCMA. The NXC-201 (formerly HBI0101) CART is provided fresh without cryopreservation.

SUMMARY:
It is a phase one study with dose escalation and safety CART in BCMA- Expressing Multiple Myeloma and AL amyloidosis Patients

DETAILED DESCRIPTION:
The intention with NXC-201 (formerly HBI0101) CART is to follow the chimeric antigen receptor T-cells (CART) approach, as for approved products, but target the B cell maturation antigen (BCMA) rather than the CD19 antigen targeted by KYMRIAHTM (tisagenlecleucel) and YESCARTATM (axicabtagene ciloleucel).

Importantly, successful results from at least three clinical trials of a BCMA targeted CAR T therapy were published (Zhao 2018, Brundo 2018, Raje 2019), with excellent results obtained for relapsed or refractory multiple myeloma (MM) patients, that validate the approach.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age

  * Voluntarily signed informed consent form (ICF)
  * Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
  * Diagnosis of MM with relapsed or refractory disease and have had at least 3 different prior lines of therapy including proteasome inhibitor, immunomodulatory therapy and at least one antibody therapy.
  * Subjects must have measurable disease, including at least one of the criteria below:

    * Serum M-protein greater or equal to 0.5 g/dL
    * Urine M-protein greater or equal to 200 mg/24 h
    * Serum free light chain (FLC) assay: involved FLC level greater or equal to 5 mg/dL (50 mg/L) provided serum FLC ratio is abnormal
    * A biopsy-proven evaluable plasmacytoma
    * Bone marrow plasma cells > 20% of total bone marrow cells
    * Non secretory patient will be allowed provided they have measurable disease by PET-CT or bone marrow aspiration, as designated.
  * Women of child-bearing potential (WCBP), must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study
  * Recovery to ≤Grade 2 or baseline of any non-hematologic toxicities due to prior treatments, excluding alopecia and Grade 3 neuropathy
  * Ability and willingness to adhere to the study visit schedule and all protocol requirements

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Determination of MTD | 21 days
  Part A: Determination of MTD Part B: Confirmation of selected dose tested (at or below MTD) ( safety )

SECONDARY OUTCOMES:
The overall survival | 2 years
  according to the IMWG Uniform Response Criteria for Multiple Myeloma
The progression-free survival | 2 years
  according to the IMWG Uniform Response Criteria for Multiple Myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Polina Stepensky, prof., Principal Investigator — Hadassah university hospital of Jerusalem
Locations (1):
- Hadassah University Hospital, Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
There will be no IPD sharing

REFERENCES:
- [Derived] Lebel E, Asherie N, Kfir-Erenfeld S, Grisariu S, Avni B, Elias S, Assayag M, Dubnikov-Sharon T, Pick M, Alexander-Shani R, Bessig N, Herr S, Shehadeh A, Ishtay A, Pimienta S, Vainstein V, Zimran E, Cohen Y, Avivi I, Cohen C, Stepensky P, Gatt ME. Efficacy and Safety of Anti-B-Cell Maturation Antigen Chimeric Antigen Receptor T-Cell for the Treatment of Relapsed and Refractory AL Amyloidosis. J Clin Oncol. 2025 Jun 10;43(17):2007-2016. doi: 10.1200/JCO-24-02252. Epub 2024 Dec 9. PMID 39653116
- [Derived] Kfir-Erenfeld S, Asherie N, Lebel E, Vainstein V, Assayag M, Dubnikov Sharon T, Grisariu S, Avni B, Elias S, Alexander-Shani R, Bessig N, Shehadeh A, Ishtay A, Zelmanovich V, Zimran E, Pick M, Roziner I, Kenett RS, Cohen Y, Avivi I, Cohen CJ, Gatt ME, Stepensky P. Clinical evaluation and determinants of response to HBI0101 (BCMA CART) therapy in relapsed/refractory multiple myeloma. Blood Adv. 2024 Aug 13;8(15):4077-4088. doi: 10.1182/bloodadvances.2024012967. PMID 38768428
- [Derived] Asherie N, Kfir-Erenfeld S, Avni B, Assayag M, Dubnikov T, Zalcman N, Lebel E, Zimran E, Shaulov A, Pick M, Cohen Y, Avivi I, Cohen C, Gatt ME, Grisariu S, Stepensky P. Development and manufacture of novel locally produced anti-BCMA CAR T cells for the treatment of relapsed/refractory multiple myeloma: results from a phase I clinical trial. Haematologica. 2023 Jul 1;108(7):1827-1839. doi: 10.3324/haematol.2022.281628. PMID 36200421
- [Derived] Kfir-Erenfeld S, Asherie N, Grisariu S, Avni B, Zimran E, Assayag M, Sharon TD, Pick M, Lebel E, Shaulov A, Cohen YC, Avivi I, Cohen CJ, Stepensky P, Gatt ME. Feasibility of a Novel Academic BCMA-CART (HBI0101) for the Treatment of Relapsed and Refractory AL Amyloidosis. Clin Cancer Res. 2022 Dec 1;28(23):5156-5166. doi: 10.1158/1078-0432.CCR-22-0637. PMID 36107221